CLINICAL TRIAL: NCT05065450
Title: Mechanisms of Amygdala-Mediated Memory Enhancement in Humans
Brief Title: Amygdala Memory Enhancement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202104033
Record Dates: First submitted 2021-08-17; First posted 2021-10-04 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Brain Diseases; Epilepsy; Memory Disorders; Traumatic Brain Injury; Cognitive Impairment; Post Traumatic Stress Disorder
MeSH Terms: conditions — Brain Diseases; Epilepsy; Memory Disorders; Brain Injuries, Traumatic; Cognitive Dysfunction; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Brain Stimulation (Experimental): Neurosurgical epilepsy patients that undergo placement of medial temporal electrode for seizure localizations will be recruited. All participants will view a series of images of emotionally-neutral objects on a computer screen. After each item presentation, they will randomly undergo either active-BLAES or sham-stimulation. Over subsequent days, free recall and recognition memory for these items, relative to new distractor items will be tested. Memory for items presented with and without stimulation will be compared. Brain activity recorded in the medial temporal lobe during item presentations will be used to predict subsequent memory. Such good and bad memory states (biomarkers) will be used to perform closed-loop stimulation when bad memory states are detected in order to enhance subsequent memory.
  Interventions: Device: Intracranial Stimulation

INTERVENTIONS:
Device: Intracranial Stimulation — Electrodes localized to the BLA will be stimulated with either active-BLAES (0.5-3.5 mA, theta-modulated gamma burst) electrical stimulation for a 1-sec duration immediately following item image presentation or sham-BLAES (zero-amplitude). At later stages of the project, stimulation parameters and timing will be varied and triggered not at random, but by real-time closed-loop analysis of memory biomarkers in the medial temporal lobe.
  Other Names: Device: ACTIVE basal lateral amygdala electrical stimulation (Active-BLAES); Device: SHAM basal lateral amygdala electrical stimulation (Sham-BLAES)

SUMMARY:
The objective is to understand how amygdala activation affects other medial temporal lobe structures to prioritize long-term memories. The project is relevant to disorders of memory and to disorders involving affect and memory, including traumatic brain injury and post-traumatic stress disorder.

DETAILED DESCRIPTION:
Direct electrical stimulation (DES) of the basolateral complex of the amygdala (BLA) can improve declarative memory, reflecting the role of the BLA in modulating memory processes in medial temporal lobe (MTL) regions as a function of emotional arousal. Thus, DES can reveal mechanisms of BLA-mediated memory enhancement relevant to human mental health and disease. DES of the BLA can be used to interrogate the function of memory circuits, especially how neuronal oscillations in the MTL support declarative memory. First, BLA is hypothesized to wield the capacity to prioritize long-term retention of information initially encountered adjacent in time over days and weeks after encoding. Second, the BLA preferentially projects to anterior MTL regions and thus is hypothesized to preferentially modulate memory processes in those anatomic regions, processes thought to support memory for non-spatial items more so than memory for spatial locations. Third, although emotional arousal, amygdala activity, MTL activity, and memory performance are typically correlated, the investigators hypothesize that DES will reveal that BLA outputs to other MTL regions cause improved memory performance by directly eliciting pro-memory oscillatory states in those networks. The expected outcomes represent a significant advancement for the basic science of normal memory function and significant movement towards novel therapeutics designed to emulate endogenous mechanisms of memory enhancement.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to understand and speak English.
* Able to provide informed consent.
* Diagnosed with epilepsy.
* Scheduled to undergo long-term intra-cranial video monitoring for seizure onset localization.
* Must be implanted with intracranial depth electrodes to the left or right amygdala, hippocampus, and parahippocampal/perirhinal cortices.

Exclusion Criteria:

* Unable to understand and speak English.
* Unable to provide informed consent.
* Not diagnosed with epilepsy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Free recall memory discriminability index (proportion recalled) | 5 years
  Proportion of items (objects, associations, and scenes) accurately recalled during the delayed recall trial will be compared with and without BLAES for each participant in a within subject design. Subsets of items may be tested after durations up to a month after initial presentation.
Recognition memory discriminability index (proportion recalled) | 5 years
  Proportion of items (objects, associations, and scenes) accurately recognized during the delayed recognition trial will be compared with and without BLAES for each participant in a within subject design. Subsets of items may be tested after durations up to a month after initial presentation.

SECONDARY OUTCOMES:
Location of single pulse evoked potential (SPEP) response to amygdala stimulation | 5 years
  Measured by presence of the evoked potential in different brain subregions (hippocampus, entorhinal cortex, perirhinal cortex, and parahippocampal cortex).
Amplitude of SPEP response to amygdala stimulation | 5 years
  Measured in microvolts.
Latency of SPEP response to amygdala stimulation | 5 years
  Measured in milliseconds.
Local field potential (LFP) of good memory state | 5 years
  Measured by relative power spectral frequency recorded at time of item presentation that predicts accurate subsequent memory performance.
LFP of bad memory state | 5 years
  Measured by relative power spectral frequency recorded at the time of item presentation that predicts inaccurate subsequent memory performance

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Inman CS, Manns JR, Bijanki KR, Bass DI, Hamann S, Drane DL, Fasano RE, Kovach CK, Gross RE, Willie JT. Direct electrical stimulation of the amygdala enhances declarative memory in humans. Proc Natl Acad Sci U S A. 2018 Jan 2;115(1):98-103. doi: 10.1073/pnas.1714058114. Epub 2017 Dec 18. PMID 29255054
- [Background] Manns JR, Bass DI. The amygdala and prioritization of declarative memories. Curr Dir Psychol Sci. 2016 Aug;25(4):261-265. doi: 10.1177/0963721416654456. PMID 27721578
- [Background] Bass DI, Manns JR. Memory-enhancing amygdala stimulation elicits gamma synchrony in the hippocampus. Behav Neurosci. 2015 Jun;129(3):244-56. doi: 10.1037/bne0000052. PMID 26030426
- [Background] Bass DI, Nizam ZG, Partain KN, Wang A, Manns JR. Amygdala-mediated enhancement of memory for specific events depends on the hippocampus. Neurobiol Learn Mem. 2014 Jan;107:37-41. doi: 10.1016/j.nlm.2013.10.020. Epub 2013 Nov 8. PMID 24211699
- [Background] Bass DI, Partain KN, Manns JR. Event-specific enhancement of memory via brief electrical stimulation to the basolateral complex of the amygdala in rats. Behav Neurosci. 2012 Feb;126(1):204-8. doi: 10.1037/a0026462. Epub 2011 Dec 5. PMID 22141467